CLINICAL TRIAL: NCT02626832
Title: Regulation of Arginine-vasopressin (AVP) in Psychiatric Disorders
Brief Title: Regulation of Arginine-vasopressin (AVP)
Acronym: REGAVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); The John B. Pierce Laboratory (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0910005875
Record Dates: First submitted 2015-11-04; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia; Depression
Keywords: vasopressin; AVP; NMDA; osmolality
MeSH Terms: conditions — Schizophrenia; Depression; Diabetes Insipidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Control (Experimental): This group is represented by healthy controls
  Interventions: Other: Procedural
- Depression (Experimental): This experimental group is represented by subjects with depression
  Interventions: Other: Procedural
- Schizophrenia (Experimental): This experimental group is represented by subjects with schizophrenia
  Interventions: Other: Procedural
- Prodromal subjects (Experimental): This experimental group is represented by subjects with prodromal symptoms for schizophrenia
  Interventions: Other: Procedural

INTERVENTIONS:
Other: Procedural — All subjects receive intravenous hypertonic saline and serial blood samples are drawn for AVP concentrations

SUMMARY:
This study aims to develop a method for the assessment of central NMDA receptor functioning in patients with depression and schizophrenia. For this purpose a transitional approach is used based on preclinical studies that show a dose-dependent relationship between the activity of hypothalamic NMDA receptor and plasma AVP response to increasing plasma osmolality. Patients with schizophrenia, depression and healthy controls participated in this study. The Investigators found that in a subgroup of patients with schizophrenia the AVP response was low and that in a subgroup of subjects with depression the AVP response was high compared to healthy controls.

DETAILED DESCRIPTION:
Evidence suggests that altered N-methyl-D-aspartate (NMDA) receptor activity and glutamate signaling may underlie the pathogenesis of both schizophrenia and depression at least in subgroups of patients. In schizophrenia, pharmacologic modeling, postmortem and imaging data suggest reduced NMDA signaling. In contrast, recent clinical trials demonstrating the efficacy of the NMDA antagonist ketamine in severely depressed patients suggest increased NMDA receptor signaling. The Investigators have conducted a proof of concept study to assess whether there is any in vivo evidence for an inverse association in depression and schizophrenia with respect to the NMDA receptor function. For this purpose the investigators used a translational approach, based on findings from animal studies that NMDA receptor is a key mediator of arginine-vasopressin (AVP) release into the bloodstream. Using hypertonic saline to induce AVP release, as done in animal studies, it was found that in a subgroup of depressed patients, NMDA receptor mediated AVP release was significantly increased, whereas in a subgroup of schizophrenia patients, the same response was abnormally low. Previous research has demonstrated that this response is well conserved. These findings are consistent with implicated NMDA receptor related abnormalities in depression and schizophrenia in subgroups of patients, and provide the first in vivo evidence towards this dichotomy.

ELIGIBILITY:
Inclusion criteria for healthy controls:

* Ages of 18-55 years from all ethnic backgrounds.
* Male or female.
* Smoker or nonsmoker.
* Written informed consent.

Exclusion criteria for healthy controls:

* DSM-IV diagnosis of psychotic, anxiety, mood disorder.
* History of major psychiatric disorder in first-degree relatives.
* A history of significant medical/neurological disease. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up (CBC with differential, SMA-7, uric acid, creatinine clearance, LFTs, TFTs, UA, Utox, Urine pregnancy test).
* A history of cardiac disease including arrhythmias; history of syncope or unexplained loss of consciousness; history of renal stones or renal failure; history of diabetes mellitus or diabetes insipidus.
* Subjects with hypertension (BP > 140/90).
* Current hyponatremia.
* Serum Ca2+ and uric acid levels that are above normal range.
* Serum creatinine outside of normal range for age.
* Creatinine clearance <70 ml/min using the Cockcroft-Gault equation (Cockcroft et al 1976) [(140-age)*(weight in kg)*(.85 if female)/(72*Cr)].
* Any medication that in the opinion of the PI could interfere with either the safety of the study and/or the outcome measures, such as diuretics of any type, lithium, carbamazepine.
* Current substance abuse/dependency determined by urine toxicology.
* Current treatment with medications with psychotropic effects.
* Current pregnancy, unsatisfactory birth control method report for females.
* IQ < 70 as determined by Wechsler Abbreviated Scale of Intelligence.
* Non-English speaking.

Inclusion criteria for patients with schizophrenia:

* Ages of 21-55 years from all ethnic backgrounds.
* Male or female.
* Smoker or nonsmoker.
* Written informed consent.
* DSM-IV diagnosis of schizophrenia or schizoaffective disorder.
* For treated patients: The patient has been on a stable dose of antipsychotics for the past month and does not require a change of medications or dose adjustment at study entry.
* For untreated patients: Has refused to be treated with medications, maintains regular clinic appointments with the clinicians, and does not pose an imminent danger to himself or others.

Exclusion criteria for patients with schizophrenia

* A history of significant medical/neurological disease. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up (CBC with differential, SMA-7, uric acid, creatinine clearance, LFTs, TFTs, UA, Utox, Urine pregnancy test).
* A history of cardiac disease including arrhythmias; history of syncope or unexplained loss of consciousness; history of renal stones or renal failure; history of diabetes mellitus or diabetes insipidus.
* Serum Ca2+ and uric acid levels that are above normal range.
* Serum creatinine outside of normal range for age.
* Creatinine clearance <70 ml/min using the Cockcroft-Gault equation [(140-age)*(weight in kg)*(.85 if female)/(72*Cr)].
* Subjects with hypertension (BP > 140/90).
* Current hyponatremia.
* Any medication that in the opinion of the PI could interfere with either the safety of the study and/or the outcome measures, such as diuretics of any type, lithium, carbamazepine.
* Currently on clozapine as clozapine may interfere with brain water regulation (Leadbetter and Shutty, 1994).
* Current substance abuse/dependency determined by urine toxicology.
* Current pregnancy, unsatisfactory birth control method report for females.
* IQ < 70 as determined by Wechsler Abbreviated Scale of Intelligence.
* Non-English speaking.

Inclusion criteria for patients with depression:

* Ages of 21-55 years from all ethnic backgrounds.
* Male or female.
* Smoker or nonsmoker.
* Written informed consent.
* DSM-IV diagnosis of major depressive disorder, unipolar.
* For treated patients: The patient has been on a stable dose of medications (antidepressants) for the past month and does not require a change of medications or dose adjustment at study entry.
* For untreated patients: Has refused to be treated with medications, maintains regular clinic appointments with the clinicians, and does not pose an imminent danger to himself or others.

Exclusion criteria for patients with depression:

* A history of significant medical/neurological disease. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up (CBC with differential, SMA-7, uric acid, creatinine clearance, LFTs, TFTs, UA, Utox, Urine pregnancy test).
* A history of cardiac disease including arrhythmias; history of syncope or unexplained loss of consciousness; history of renal stones or renal failure; history of diabetes mellitus or diabetes insipidus.
* Serum Ca2+ and uric acid levels that are above normal range.
* Serum creatinine outside of normal range for age.
* Creatinine clearance <70 ml/min using the Cockcroft-Gault equation [(140-age)*(weight in kg)*(.85 if female)/(72*Cr)].
* Subjects with hypertension (BP > 140/90).
* Current hyponatremia.
* Any medication that in the opinion of the PI could interfere with either the safety of the study and/or the outcome measures, such as diuretics of any type, lithium, carbamazepine.
* Current substance abuse/dependency determined by urine toxicology.
* Current pregnancy, unsatisfactory birth control method report for females.
* IQ < 70 as determined by Wechsler Abbreviated Scale of Intelligence.
* Non-English speaking.

Inclusion criteria for patients from the PRIME Clinic:

* Ages of 18-40 years from all ethnic backgrounds.
* Male or female.
* Smoker or nonsmoker.
* Written informed consent.

Exclusion criteria for patients from the PRIME Clinic:

* A history of significant medical/neurological disease. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up (CBC with differential, SMA-7, uric acid, creatinine clearance, LFTs, TFTs, UA, Utox, Urine pregnancy test).
* A history of cardiac disease including arrhythmias; history of syncope or unexplained loss of consciousness; history of renal stones or renal failure; history of diabetes mellitus or diabetes insipidus.
* Serum Ca2+ and uric acid levels that are above normal range.
* Serum creatinine outside of normal range for age.
* Creatinine clearance <70 ml/min using the Cockcroft-Gault equation [(140-age)*(weight in kg)*(.85 if female)/(72*Cr)].
* Subjects with hypertension (BP > 140/90).
* Current hyponatremia.
* Any medication that in the opinion of the PI could interfere with either the safety of the study and/or the outcome measures, such as diuretics of any type, lithium, carbamazepine.
* Currently on clozapine as clozapine may interfere with brain water regulation (Leadbetter and Shutty, 1994).
* Current substance abuse/dependency determined by urine toxicology.
* Current pregnancy, unsatisfactory birth control method report for females.
* IQ < 70 as determined by Wechsler Abbreviated Scale of Intelligence.
* Non-English speaking.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-02; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AVP response to plasma osmolality as measured by slopes between the two variables | Within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Handan Gunduz-Bruce, MD, MBA, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - The John Pierce Laboratory, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut